CLINICAL TRIAL: NCT00321386
Title: Parameters for Disease Progression in Chinese Patients With Normal Tension Glaucoma
Brief Title: Analysis of Clinical Profiles of Chinese Patients With Normal Tension Glaucoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Hong Kong Eye Hospital (Other); Prince of Wales Hospital, Shatin, Hong Kong (Other)
Responsible Party: Dr. Dexter Leung/ Honorary Clinical Assistant Professor, Department of Ophthalmology & Visual Sciences, The Chinese University of HK
Other Study IDs: KC/KE 05-0169/ER-1; CRE-2005.434
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Glaucoma
Keywords: Glaucoma; Open Angle; Normal Tension
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood taking for glaucoma genetics analysis shall be performed.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To obtain demographic and baseline ophthalmic parameters (such as Intraocular Pressure profiles, disc morphological characteristics, central corneal thickness, peripapillary retinal nerve fibre layer thickness and its serial changes, visual field changes, severity of any medical associations-e.g. hypertension, migraine, strokes, silent cerebral infarcts) with non-invasive measurements, in Chinese Patients with Normal Tension Glaucoma

DETAILED DESCRIPTION:
This is a multi-centered non-interventional descriptive study. The Declaration of Helsinki is followed. All procedures will be conducted in accordance with the GCP guidelines.

About 100 Consecutive NTG glaucoma patients will be included in this study. NTG is defined as:

1. Six median untreated intraocular pressure consistently less than 21 mm Hg, with no more than 1 reading = 23 mmHg or 24 mmHg, and with no single measurement greater than 24 mm Hg,
2. Open drainage angles on gonioscopy,
3. Typical optic disc damage with glaucomatous cupping and loss of neuroretinal rim,
4. Absence of any secondary cause for a glaucomatous optic neuropathy (trauma, steroids, uveitis),
5. Glaucomatous visual field defect compatible with glaucomatous optic neuropathy.

Age and sex-matched normal control subjects and age, sex, severity-matched POAG control subjects will be recruited.

Randomization not required as this will be a non-interventional descriptive study.

A complete baseline ophthalmic assessment will be performed with Snellen visual acuity (VA), Best-corrected VA, intraocular pressure (IOP) measurements, slit lamp examination, gonioscopy, disc assessment and dilated fundal examination.

These measurements were performed at recruitment and then at 3,6,9,12 months after the intervention. The details of some of these measurements were as follows.

All IOP was measured with Goldmann applanation tonometry. The median of 5 readings were taken. Gonioscopy was carried out first using a Goldmann 2-mirror gonioscope. The examination was carried out at the lowest level of illumination that permitted a view of the angle and at high magnification (×16 to ×25). A 1-mm light beam was reduced to a very narrow slit, and was offset horizontally for assessing superior and inferior angles and vertically for nasal and temporal angles. Care was taken to avoid light falling on the pupil during gonioscopy. Slight tilting to gain a view over the convexity of the iris was permitted, but further manipulation of the lens or redirection of gaze was avoided because of the possibility of exerting pressure on the cornea and artificially widening the angle. The drainage angle was graded according to Shaffer's convention in each quadrant. The average angle width was calculated by adding the Shaffer grade in each quadrant and dividing by 4. Indentation gonioscopy using a Posner lens was also used to detect PAS, and the number of clock hours of PAS was recorded. All gonioscopy was performed by a single investigator for standardization.

The vertical CDR was taken to be the longest vertical cup diameter divided by the longest vertical disc diameter. Estimates were made to the nearest 0.05. The vertical disc diameter was examined. All features of a glaucomatous optic neuropathy were noted.

All subjects underwent static automated white-on-white threshold perimetry (program 24- 2, SITA standard, model 750, Humphrey Instruments, Dublin, CA), and the first reliable VF was used in our analysis. The global indices mean deviation (MD), and pattern standard deviation (PSD) were documented for all cases. After finding the proportion of VF that is reliable, the VF was then scored using the tested scoring algorithm developed for the Advanced Glaucoma Intervention Study (AGIS).

Minimal criteria for glaucomatous VF defect were as follows: glaucoma hemifield test outside normal limits, pattern standard deviation with a P value of <5%, or a cluster of ≥3 points in the pattern deviation plot in a single hemifield (superior or inferior) with P value of <5%, one of which must have a P value of <1%. Any one of the preceding criteria, if repeatable, was considered sufficient evidence of a glaucomatous VF defect.

Subjects will be verified by diurnal tension curve, which was recorded no more than one year before inclusion in the present study.

Systemic haemodynamics Systolic, diastolic, and mean blood pressures (SBP, DBP, MAP) were measured on the upper arm by an automated oscillometric device. Pulse rate (PR) and blood oxygenation was automatically recorded from a finger pulse oximetric device (HP-CMS patient monitor, Hewlett Packard, Palo Alto, CA, USA).

Measurement of intraocular pressure (IOP) A Median of 3 readings for each subject with Goldmann applanation tonometer was used for each measurement of intraocular pressure.

Fundus Photography and Optical Coherence Tomography (OCT) A baseline fundus photo will be performed for all participants. A baseline OCT for retinal nerve fiber layer thickness and optic nerve head parameters will be determined. Serial changes of these parameters will be correlated to VF indices.

Dynamic Contour Tonometry (DCT) and Ocular Response Analyzer (ORA) will also be performed on these subjects.

A history of the following systemic conditions was recorded: systemic hypertension (HT), hypotension, ischemic heart disease (IHD), arrhythmia, diabetes mellitus (DM), hypercholesterolemia, cerebral vascular accidents (CVA), migraine, obstructive sleep apnea (OSA), sensorineural hearing loss and Raynaud's phenomenon. All diagnoses were obtained from the history and confirmed by the clinical management system of the Hong Kong Hospital Authority, which is a computerized database connecting all public hospitals and clinics in Hong Kong.

Systemic use of statins, beta-blockers, angiotensin-converting-enzyme-inhibitors (ACEI), calcium-channel-blockers, aspirin and diuretics was also noted.

ELIGIBILITY:
Inclusion Criteria:

* All Chinese patients with age>18 years old with Normal Tension Glaucoma will be recruited

Exclusion Criteria:

* Diseases that precluded accurate measurement of IOP, visual acuity, retinal nerve fiber layer thickness, and visual field tests.
* Previous ocular surgery per se is not an exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Normal Tension Glaucoma recruited from a teritary University Eye Hospital setting.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2003-12; Primary Completion 2008-12 (Actual); Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: LEUNG YL Dexter, MBChB, FRCS, Principal Investigator — Glaucoma Service, Hong Kong Eye Hospital; LAM SC Dennis, MD, FRCOphth, Study Chair — Chinese University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Hong Kong Eye Hospital, Hong Kong
  - Prince of Wales Hospital, Hong Kong

REFERENCES:
- [Background] Drance S, Anderson DR, Schulzer M; Collaborative Normal-Tension Glaucoma Study Group. Risk factors for progression of visual field abnormalities in normal-tension glaucoma. Am J Ophthalmol. 2001 Jun;131(6):699-708. doi: 10.1016/s0002-9394(01)00964-3. PMID 11384564
- [Result] Leung DY, Tham CC, Li FC, Kwong YY, Chi SC, Lam DS. Silent cerebral infarct and visual field progression in newly diagnosed normal-tension glaucoma: a cohort study. Ophthalmology. 2009 Jul;116(7):1250-6. doi: 10.1016/j.ophtha.2009.02.003. Epub 2009 May 30. PMID 19481813
- [Result] Leung DY, Li FC, Kwong YY, Tham CC, Chi SC, Lam DS. Simvastatin and disease stabilization in normal tension glaucoma: a cohort study. Ophthalmology. 2010 Mar;117(3):471-6. doi: 10.1016/j.ophtha.2009.08.016. Epub 2010 Jan 4. PMID 20045568
- [Result] Leung DY, Kwong YY, Li FC, Tham CC, Chi SC, Lam DS. Comparison of the clinical characteristics of normal tension glaucoma patients with pretreatment intraocular pressures in the high-teens and low-teens. Br J Ophthalmol. 2010 May;94(5):663-5. doi: 10.1136/bjo.2009.163014. No abstract available. PMID 20447973
- [Derived] Leung DY, Iliev ME, Chan P, Baig N, Chi SC, Tham CC, Lam DS. Pressure-cornea-vascular index (PCVI) for predicting disease progression in normal tension glaucoma. Br J Ophthalmol. 2011 Aug;95(8):1106-10. doi: 10.1136/bjo.2009.175992. Epub 2010 Aug 7. PMID 20693562